CLINICAL TRIAL: NCT02678429
Title: Atlas Predicted DBS Settings in Essential Tremor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to fully enroll no data analysis planned
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Fenna Phibbs, Assistant Professor of Neurology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 160155
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBS programming, standard of care (Active Comparator): DBS settings determined from the standard Neurologist symptomatic response first then change to settings from Atlas
  Interventions: Device: Change DBS programming
- DBS progamming from Atlas (Experimental): DBS settings determined from the a functional atlas first then change to settings determined by standard of care
  Interventions: Device: Change DBS programming

INTERVENTIONS:
Device: Change DBS programming — Patient will change their DBS settings to move from one DBS setting to the other, allowed one hour to adjust to the new setting prior to testing

SUMMARY:
Programming Deep Brain Stimulation for the treatment of Essential Tremor can be a time intensive process. Using an atlas created using functional tremor responses in the operating room to determine the optimal settings would lead to a faster response for the patient and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

Seleced for DBS of the VIM nucleus at Vanderbilt Medical center Diagnosis of essential tremor

Exclusion Criteria:

Unable to use the patient handheld programmer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DBS Programming, Standard of Care: DBS settings determined from the standard Neurologist symptomatic response, first
  Change DBS programming: Patient will change thier settings to move from one group to the other to trial the other DBS settings
- DBS Progamming From Atlas: DBS settings determined from the a functional atlas only,first
  Change DBS programming: Patient will change thier settings to move from one group to the other to trial the other DBS settings
Period: Overall Study
Arm/Group | DBS Programming, Standard of Care | DBS Progamming From Atlas
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBS Programming, Standard of Care | DBS Progamming From Atlas | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Fahn-Tolusa-Marsden Tremor Rating Scale
Description: Tremor quantification
Time Frame: 1 month
Population: Data analysis was not completed because only one participant completed the DBS Programming from Atlas arm and disclosing data could violate privacy interests.
Arm/Group | DBS Programming, Standard of Care | DBS Progamming From Atlas
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | DBS Programming, Standard of Care | DBS Progamming From Atlas
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

LIMITATIONS AND CAVEATS:
Unable to fully recruit for the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT02678429/Prot_SAP_000.pdf